CLINICAL TRIAL: NCT03532854
Title: A Randomized, Open-label, Multiple-dose, Crossover Clinical Trial to Evaluate the Safety/Tolerability and Pharmacokinetic Drug-drug Interaction Between LGEV1801 and LGEV1802 in Healthy Korean Male Volunteers
Brief Title: Evaluating a Pharmacokinetic Drug Interaction Between LGEV1801 and LGEV1802
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LG-EVCL001
Record Dates: First submitted 2018-05-08; First posted 2018-05-22 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Healthy Male Volunteers
MeSH Terms: interventions — Valsartan; Ezetimibe; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence A (Experimental): Ezetimibe/Rosuvastatin -> Valsartan -> Valsartan and Ezetimibe/Rosuvastatin
  Interventions: Drug: Valsartan; Drug: Ezetimibe/Rosuvastatin
- Sequence B (Experimental): Valsartan -> Valsartan and Ezetimibe/Rosuvastatin-> Ezetimibe/Rosuvastatin
  Interventions: Drug: Valsartan; Drug: Ezetimibe/Rosuvastatin
- Sequence C (Experimental): Valsartan and Ezetimibe/Rosuvastatin -> Ezetimibe/Rosuvastatin -> Valsartan
  Interventions: Drug: Valsartan; Drug: Ezetimibe/Rosuvastatin
- Sequence D (Experimental): Ezetimibe/Rosuvastatin -> Valsartan and Ezetimibe/Rosuvastatin-> Valsartan
  Interventions: Drug: Valsartan; Drug: Ezetimibe/Rosuvastatin
- Sequence E (Experimental): Valsartan -> Ezetimibe/Rosuvastatin -> Valsartan and Ezetimibe/Rosuvastatin
  Interventions: Drug: Valsartan; Drug: Ezetimibe/Rosuvastatin
- Sequence F (Experimental): Valsartan and Ezetimibe/Rosuvastatin -> Valsartan -> Ezetimibe/Rosuvastatin
  Interventions: Drug: Valsartan; Drug: Ezetimibe/Rosuvastatin

INTERVENTIONS:
Drug: Valsartan — Valsartan P.O
  Other Names: Diovan
Drug: Ezetimibe/Rosuvastatin — Ezetimibe/Rosuvastatin P.O
  Other Names: Rosuzet

SUMMARY:
The purpose of this study is to evaluate the drug-drug interaction between LGEV1801 and LGEV1802 in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male
* Age between 19 and 50
* Subjects with BMI of 18~27 kg/m2 with a weight of 55kg or more
* Subjects with SBP of 90~150 mmHg and DBP of 60~150 mmHg
* Signed informed consent

Exclusion Criteria:

* Presence of medical history or a concurrent disease
* Has a history of hypersensitivity to IP ingredients

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2018-08-25 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
AUCT,ss | Day 1~Day 8
Cmax,ss | Day 1~ Day 8

CONTACTS AND LOCATIONS:
Locations (1):
- LG chem, Seoul, Gangseo-Gu, South Korea

IPD SHARING:
Plan to Share IPD: No